CLINICAL TRIAL: NCT03854643
Title: Influence of the Pilates Method in the Treatment of Unexpected Chronic Lombar Pain: Clinical Controlled, Randomized and Double Clinical Test.
Brief Title: Influence of the Pilates Method in the Treatment of Unexpected Chronic Lombar Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cruzeiro do Sul (Other)
Responsible Party: Principal Investigator, Leandro Lazzareschi, Principal Investigator, University of Mogi das Cruzes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90158318.3.0000.5497
Record Dates: First submitted 2019-02-16; First posted 2019-02-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lower Back Pain
Keywords: pilates method
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blind researcher will be responsible for evaluating the volunteers. It is worth mentioning that this researcher will not have access to the research group that the participants will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates group (Experimental): 17 (seventeen) volunteers of both genders, aged between 18 and 35 years, were recruited for at least 3 (three) months with non-specific back pain. Pilates exercises were performed three times a week for 4 weeks, totaling 12 treatment sessions. Each session lasted 40 minutes and was performed by a researcher with training in the method and previous training in the exercise. The patients were evaluated as follows: initial assessment, after two weeks, after four weeks and a follow up after three months.
  Interventions: Other: Pilates group
- Control group (Experimental): 17 (seventeen) volunteers of both genders, aged between 18 and 35 years, were recruited for at least 3 (three) months with non-specific back pain. These patients did not receive any type of intervention. The patients were evaluated as follows: initial assessment, after two weeks, after four weeks and a follow up after three months.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Pilates group — Pilates exercises were performed three times a week for 4 weeks, totaling 12 treatment sessions. Each session lasted 40 minutes and was performed by a researcher with training in the method and previous training in the exercise. The patients were evaluated as follows: initial assessment, after two weeks, after four weeks and a follow up after three months.
  Arms: Pilates group
Other: Control group — These patients did not receive any type of intervention. The patients were evaluated as follows: initial assessment, after two weeks, after four weeks and a follow up after three months.
  Arms: Control group

SUMMARY:
This study aims to verify the influence of the Pilates Method on the improvement of pain in patients with non-specific chronic low back pain

DETAILED DESCRIPTION:
Nonspecific low back pain is defined as localized pain and discomfort between the lower margins of the costal gradis and the lower gluteal folds. Chronic low back pain may be associated with central sensitization (CS) which is a proposed physiological phenomenon in which a deregulation in the central nervous system. Another relevant point related to worsening pain is kinesiophobia, which is fear of movement due to pain which impedes the movement or causes the person to gradually decrease their activities, thus limiting their functions, and restricting their participation in activities of daily living. The research design is a randomized, controlled, blinded clinical trial on the influence of central stabilization on the basis of the Pilates method in improving pain, kinesiophobia, central sensitization and function in patients with chronic low back pain of non-specific origin. It is a research with four evaluations: pre-treatment, post-two weeks, post four weeks and three months after the end of treatment. An evaluation form will be used, containing questions about personal data, history of diseases, ethylism, smoking, medications used and pain intensity by the numerical scale of pain. The Tampa scale for kinesiophobia will also be used. The Central Sensitization questionnaire, which has two parts, part A containing 25 questions about the presence of pain in the last 3 months and part B containing 10 questions about possible medical diagnoses will be used. Finally, the Oswestry 2.0 Disability Index will be applied. 34 (thirty-four) volunteers, of both genders, aged between 18 and 35 years old will be recruited for at least 3 (three) months of non-specific back pain; of which 17 (seventeen) will undergo the Pilates Method and 17 (seventeen) will be part of the control group. Pilates exercises will be performed three times a week for 4 weeks, totaling 12 sessions of treatment, by a researcher with training in the method and previous training in performing the exercises. The re-evaluations will be performed after the sixth treatment session (Pilates group) and two weeks after the initial evaluation (control group), after the twelfth session (Pilates group) and after four weeks for the control group. A reevaluation will also be performed after 3 months of treatment, in order to analyze how well the Pilates method was effective in maintaining the improvement of the patient's clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Present lumbar pain of degree greater than or equal to 3;
* Present lumbar pain for twelve weeks or more;
* Present low back pain without it being related to any specific pathology or cause;
* The Volunteers may not be undergoing physiotherapeutic or drug treatment

Exclusion Criteria:

* Volunteers who present with pain grade 1 or 2 of low back pain;
* Volunteers with severe movement limitations;
* Neurological or neurological diseases that interfere with significant neuromotor
* Individuals who did not agree to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 34 (thirty-four) volunteers of both genders, aged between 18 and 35 years with non-specific back pain complaint for at least three (3) months
Enrollment: 34 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
lower back pain | 3 months
  Intensity of pain through the visual analogic scale, which contains 11 points, ranging from 0 to 10, with 0 corresponding to "no pain" and 10 to unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Institute of Health, Mogi das Cruzes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No